CLINICAL TRIAL: NCT07137962
Title: Comparison Between Pericapsular Nerve Group Block Versus Fascia Iliaca Compartment Block Versus Caudal Block for Postoperative Analgesia in Hip Surgeries in Children, A Randomized Controlled Clinical Trial
Brief Title: Pericapsular Nerve Group Block vs. Fascia Iliaca Compartment Block vs. Caudal Block for Hip Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nagy Malak , MD, Lecturer of anesthesia ,SICU and pain, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS-441- 2024
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Regional Anesthesia Morbidity; Hip Surgeries; Perioperative Analgesia
Keywords: PENG block; Caudal block; FICB; Pediatrics; Hip Surgeries

STUDY DESIGN:
Intervention Model Description: Nerve blocks were performed following anesthesia induction and before initiation of surgery, the patient was placed in a supine position according to study group include PENG Block, FICB and caudal Block.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Computer-generated randomization numbers were used for random allocation and each patients' code was kept in an opaque sealed envelope. Patients were randomly allocated with 1:1:1 allocation ratio into three groups in a parallel manner.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: PENG Block (Active Comparator): The curvilinear low-frequency (2-5 MHz) ultrasound probe was placed over the line parallel to the inguinal ligament. It was subsequently rotated 45° to identify the anterior inferior iliac spine, the ilio-pubic eminence, and the psoas tendon. A needle was inserted in the plane to place the tip in the musculo-fascial plane between the pubic ramus posteriorly and the psoas tendon anteriorly, using the hydro-dissection technique. Following negative aspiration, a total volume of 0.5 ml/kg of 0.25% bupivacaine was injected.
  Interventions: Procedure: PENG Block
- Group B: FICB block (Active Comparator): The linear ultrasound probe was placed over the inguinal ligament in the sagittal plane, inferomedial to the anterior superior iliac spine. Upon identifying the "bow-tie sign" formed by the sartorius muscle and the internal oblique muscle by sliding medially and rotating the probe. 22-gauge echogenic needle was introduced 1 cm cephalad to the inguinal ligament to place the needle tip in the space between the internal oblique and iliacus muscles, using the hydro-dissection technique. A total volume of 0.5 mL/kg of bupivacaine 0.25% was injected following negative aspiration.
  Interventions: Procedure: FICB Block
- Group C:Caudal Block (Active Comparator): The patient was placed in the left lateral position with the upper hip flexed at 90° and the lower hip flexed at 45°. The region was then swabbed in a craniocaudal direction with 70% alcohol. After palpating the landmarks (the upper posterior iliac spine and sacral hiatus from the edges of an equilateral triangle), an epidural puncture was performed in the most proximal region of the sacral hiatus with the needle inclined 45-60° to the skin. While palpating with the index finger of the left hand, a needle was inserted immediately below the spinous process S4. After perforating the membrane, which occludes the sacral hiatus, the needle was advanced no more than 1-3 mm to avoid a bloody puncture or an intrathecal injection. Bupivacaine 0.25% at a dose of 1 ml/kg was injected, with care taken to not exceed the maximum recommended dose (2 mg/kg).
  Interventions: Procedure: Caudal Block

INTERVENTIONS:
Procedure: PENG Block — The curvilinear low-frequency (2-5 MHz) ultrasound probe was placed over the line parallel to the inguinal ligament. It was subsequently rotated 45° to identify the anterior inferior iliac spine, the ilio-pubic eminence, and the psoas tendon.
  A 22-gauge echogenic needle was inserted in plain to place the tip in musculo-fascial plain between pubic ramus posteriorly and psoas tendon anteriorly, using hydro-dissection technique. Following negative aspiration, a total volume of 0.5 ml/kg of 0.25% bupivacaine was injected.
  Arms: Group A: PENG Block
Procedure: FICB Block — The linear ultrasound probe was placed over the inguinal ligament in the sagittal plane, inferomedial to the anterior superior iliac spine. Upon identifying the "bow-tie sign" formed by the sartorius muscle and the internal oblique muscle by sliding medially and rotating the probe. 22-gauge echogenic needle was introduced 1 cm cephalad to the inguinal ligament to place the needle tip in the space between the internal oblique and iliacus muscles, using the hydro-dissection technique. A total volume of 0.5 mL/kg of bupivacaine 0.25% was injected following negative aspiration.
  Arms: Group B: FICB block
Procedure: Caudal Block — After induction of general anesthesia, the patient was placed in the left lateral position with the upper hip flexed at 90° and the lower hip flexed at 45°. The region was then swabbed in a craniocaudal direction with a 70% alcohol solution.
  After palpating the landmarks (the upper posterior iliac spine and sacral hiatus from the edges of an equilateral triangle), an epidural puncture was performed in the most proximal region of the sacral hiatus with the needle inclined 45-60° to the skin. While palpating with the index finger of the left hand, a needle was inserted immediately below the spinous process S4. After perforating the membrane, which occludes the sacral hiatus, the needle was advanced no more than 1-3 mm to avoid a bloody puncture or an intrathecal injection. Bupivacaine 0.25% at a dose of 1 ml/kg was injected.
  Arms: Group C:Caudal Block

SUMMARY:
The study aims to compare the effect of pericapsular nerve group block versus fascia iliaca compartment block versus caudal block regarding Postoperative analgesia in children undergoing hip surgeries.

DETAILED DESCRIPTION:
Study included ASA I, II,1-6 years old from both sexes, scheduled for elective hip surgery.while exclusion criteria include ASA III and IV, Allergy to any medication used, neurological or psychological disorders, anatomic abnormalities or infection at site of injection and bleeding disorders (international normalized ratio (INR) >1.5 and/or platelet count <100,000/µL).

Computer-generated randomization numbers were used for random allocation and each patients' code was kept in an opaque sealed envelope. Patients were randomly allocated with 1:1:1 allocation ratio into three groups in a parallel manner:

Group A: patients received pericapsular nerve block group (PENG) block with 0.25% bupivacaine 0.5 ml/kg.

Group B: patients received fascia iliaca compartment block (FICB) with 0.25% bupivacaine 0.5 ml/kg.

Group C: patients received caudal block with 0.25% bupivacaine 1 ml/kg. On the day before the surgery, pre-operative assessment was performed, Medical and surgical history were taken, examination (airway to exclude difficult airway, chest, back, abdomen, and limbs to exclude infection at injection site and anatomical deformities) was performed.

Standard monitoring devices such as ECG, non-invasive blood pressure, pulse oximeter, and capnography were applied. Baseline blood pressure and heart rate were recorded.

General anesthesia was induced using inhalational induction with 8% sevoflurane and 50% oxygen administered via a face mask. intravenous cannula 20G was subsequently placed. fentanyl (1 mcg/kg) was given. Intubation was facilitated by atracurium (0.5 mg/kg), and then an appropriately sized endotracheal tube was placed.

All patients were mechanically ventilated with a targeted Et CO2 of 30-35 mmHg. Anesthesia was maintained with Isoflurane 1.2 % (1 MAC) to 1.5 %, depending on hemodynamics of the patient) in a mixture of 50% air and oxygen throughout the procedure. Another IV cannula was secured as per our standard protocol.

Intraoperative hypothermia was prevented by operating table mattress or operating room heater and warm intravenous fluids (15 mL/kg lactated ringer solution in the first hour, then completed according to the 4: 2: 1 rule: 4 mL/kg/h for the first 10 kg of weight, 2 mL/kg/h for the second 10 kg, and 1 mL/kg/h for each remaining kilogram). Replacement of losses: blood loss was replaced by non-glucose crystalloids in a ratio of 3: 1. It was replaced by packed RBCs guided by serum hemoglobin.

Nerve blocks were performed following anesthesia induction and before initiation of surgery, the patient was placed in a supine position, The region was then swabbed in a craniocaudal direction with a 70% alcohol solution. Intensive disinfection with alcoholic solution, sterile drapes, and the use of sterile gloves is standard for all regional blockades, all blocks were performed by an experienced anesthesiologist who was otherwise not involved in the study. The ultrasound machine used Sonosite S-Nerve Ultrasound System with linear probe, frequency: 6-15 MHz.

PENG Block:

The curvilinear low-frequency (2-5 MHz) ultrasound probe was placed over the line parallel to the inguinal ligament. It was subsequently rotated 45° to identify the anterior inferior iliac spine, the ilio-pubic eminence, and the psoas tendon.

A 22-gauge echogenic needle was inserted in plain to place the tip in musculo-fascial plain between pubic ramus posteriorly and psoas tendon anteriorly, using hydro-dissection technique. Following negative aspiration, a total volume of 0.5 ml/kg of 0.25% bupivacaine was injected.

FICB block:

The linear ultrasound probe was placed over the inguinal ligament in the sagittal plane, inferomedial to the anterior superior iliac spine. Upon identifying the "bow-tie sign" formed by the sartorius muscle and the internal oblique muscle by sliding medially and rotating the probe. 22-gauge echogenic needle was introduced 1 cm cephalad to the inguinal ligament to place the needle tip in the space between the internal oblique and iliacus muscles, using the hydro-dissection technique. A total volume of 0.5 mL/kg of bupivacaine 0.25% was injected following negative aspiration.

Caudal Block:

After induction of general anesthesia, the patient was placed in the left lateral position with the upper hip flexed at 90° and the lower hip flexed at 45°. The region was then swabbed in a craniocaudal direction with a 70% alcohol solution. Intensive disinfection with alcoholic solution, sterile drapes, and the use of sterile gloves is standard for all neuraxial blockades at our institution.

After palpating the landmarks (the upper posterior iliac spine and sacral hiatus from the edges of an equilateral triangle), an epidural puncture was performed in the most proximal region of the sacral hiatus with the needle inclined 45-60° to the skin. While palpating with the index finger of the left hand, needle was inserted immediately below the spinous process S4. After perforating the membrane, which occludes the sacral hiatus, the needle was advanced no more than 1-3 mm to avoid a bloody puncture or an intrathecal injection. Bupivacaine 0.25% at a dose of 1 ml/kg was injected, with care taken to not to exceed the maximum recommended dose (2 mg/kg).

In all groups, hemodynamic parameters (non-invasive arterial blood pressure (mean, systolic, and diastolic), heart rate, and oxygen saturation) were recorded at baseline, 5 minutes after intubation, and every 10 minutes till the end of the surgery. Skin incisions were allowed 10 minutes after performing the block.

Failed blocks (increase in HR and mean arterial pressure (MAP) >20% from the baseline with skin incision) were treated with 1 mcg/kg of fentanyl. Patients with failed block were excluded from the study.

If hypotension occurred (defined as a decrease in mean arterial pressure (MAP) >30% from baseline value), patients were treated with 0.3 - 1.2 mg / kg ephedrine until hypotension is resolved. If bradycardia occurred (defined as a decrease in HR > 30% from baseline readings), it was treated with atropine 0.02 mg/kg IV.

After skin closure, inhalational anesthesia was discontinued, and reversal of muscle relaxation was achieved with atropine (0.02 mg/kg) and neostigmine (0.05 mg/kg).

after the return of the patient's spontaneous breathing. The patient was extubated fully awake (opening the eyes). Patients were then transferred to the post-anesthesia care unit (PACU) for 60 minutes for monitoring.

In PACU, vital signs (heart rate, arterial blood pressure, and oxygen saturation) were assessed every 10 minutes. After discharging the patient from the PACU, the analgesic plan was IV paracetamol (15 mg/kg) every 8 hours.

Face, Legs, Activity, Cry, and Consolability (FLACC) pain scale was recorded every 2 h in the first 8 h, then every 4 h till 24 h postoperative. Rescue analgesia is in the form of IV morphine 0.05 mg/kg was given as rescue analgesia if the FLACC Score was ≥ 4 (Table 1) (26).

Maximal daily morphine didn't exceed 0.3 mg/kg. Time to first rescue analgesia was recorded.

Measurement Data : Patient's characteristics include age in years, weight in kilograms, gender, and type of surgery, Hemodynamic parameters (non-invasive arterial blood pressure, heart rate, and oxygen saturation) were recorded at baseline, 5 minutes after intubation, every 10 minutes till the end of the surgery, immediately after extubation, and every 10 minutes in PACU for 1 hour till the discharge of the patient, Total opioid consumption in the first 24 hours postoperative., FLACC Pain Scale every 2 h in the first 8 h, then every 4 h till 24 h postoperative, Time for first rescue analgesia in the first 24 hours postoperative ,Intraoperative total opioid consumption, Incidence of postoperative nausea and vomiting in the first 24 hours and Incidence of complications (bradycardia, hypotension, respiratory depression)

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II,1-6 years old from both sexes, scheduled for elective hip surgery.

Exclusion Criteria:

* ASA III and IV, Allergy to any medication used, neurological or psychological disorders, anatomic abnormalities or infection at site of injection and bleeding disorders (international normalized ratio (INR) >1.5 and/or platelet count <100,000/µL).

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption | The first 24 hours postoperative.
  Total opioid (morphine) (mg) consumption in the first 24 hours postoperative.

SECONDARY OUTCOMES:
FLACC Pain Scale | 24 hours
  FLACC Pain Scale every 2 h in the first 8 h, then every 4 h till 24 h postoperative,
Time for first rescue analgesia | 24 hours
  Time (hr) for first rescue analgesia in the first 24 hours post-operative
Total opioid consumption | time of operation up to 6 hours
  Intra-operative total opioid (fentanyl) (mcg/kg) consumption
Postoperative nausea and vomiting | 24 hours
  Incidence of postoperative nausea and vomiting in first 24 hours
Incidence of complications | 24 hours
  Incidence of complications (bradycardia, hypotension, respiratory depression as bradypnea or hypoxia in PACU).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university Hospitals. kasralainy, Cairo, Egypt